CLINICAL TRIAL: NCT01465880
Title: A Single-centre, Dose Titration Study in Healthy Volunteers (Smokers and Non-smokers) to Evaluate the Capacity of 2-cyanoethylmercapturic Acid (CEMA) to Detect Low Level of Cigarette Smoking Exposure
Brief Title: Smoking Research Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PIPA_CEMA_01
Record Dates: First submitted 2011-10-14; First posted 2011-11-07 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Smoking; Non-smoking
Keywords: Smoking research study
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part B. Healthy Caucasian adult non-smokers (No Intervention): Non-smokers
- Part A.Healthy Caucasian adult smokers (Experimental): No product will be investigated in this study. Smokers will smoke their own conventional cigarettes only.
  Interventions: Other: Part A

INTERVENTIONS:
Other: Part A — Smoking abstinence, smoking 2 and 4 cigarettes
  Arms: Part A.Healthy Caucasian adult smokers

SUMMARY:
The purpose of this study is to develop a fit-for-purpose biochemical verification tool that can be used to detect concomitant use of a few (less than 5) conventional cigarettes.

DETAILED DESCRIPTION:
This study will be performed in two parts. The first part, Part A, is a dose titration study in healthy smokers with incremental cigarette consumption performed in confinement. The second part, Part B, is an observational study on healthy non-smokers in an ambulatory setting

PART A (smokers only)

A screening visit will be conducted within 4 weeks prior to admission to the investigational site. The 8-day confinement period consists of the admission day (Day1), 1 day ad-libitum smoking (Day0), 3 days of smoking abstinence (Day1-3), 2-day exposure period smoking 2 and 4 cigarettes (Day4-5), and the day of discharge (Day6) followed by a 7-day safety follow-up period. Urine collection will be performed for each subject from Day0 to Day5 in 4 intervals.

PART B (non-smokers)

Screening visit will be conducted within 4 weeks prior to the ambulatory Visit 1 (collection of 24-hour urine and spot urine) to the investigational site. The minimum interval between the screening and Visit 1 is of 7 days.

ELIGIBILITY:
Inclusion Criteria:

Common criteria to smokers and non-smokers

1. Subject is able to understand the information provided in the Subject Information sheet and Informed Consent Form (ICF)
2. Subject has signed the ICF
3. Subject of Caucasian origin
4. Aged from 23 to 55 years
5. Having acceptable health conditions as judged by the Investigator at the screening visit based on clinical laboratory parameters (clinical biochemistry, urine analysis and standard haematology), spirometry, serology, urine drug screen, vital signs, physical examination, ECG, and medical history

   Specific to smokers
6. Current smoker based on self-reporting who smoke 5 to 15 commercially available non-mentholated conventional cigarettes (no brand restrictions) with a maximum tar yield of 10 mg (ISO method, as labelled on the cigarette package) smoking at least for the last 3 consecutive years. The smoking status will be verified at screening based on a urinary cotinine test (cotinine ≥200ng/ml)
7. Subject is willing to smoke according to the smoking regimen of the study

   Specific to non-smokers
8. Non-smoker based on self-reporting who have not used any tobacco or nicotine containing product including commercially available cigarettes, hand-rolled cigarettes, cigars, pipes, snuff, electronic cigarettes, similar devices, and nicotine replacement therapy within the last 12 months. The non-smoking status of the subject will be verified at screening based on a urinary cotinine test (cotinine <200ng/ml)

Exclusion Criteria:

Common criteria to smokers and non-smokers

1. As per judgement of the Investigator, any subject who cannot participate in the study for any reason (e.g., medical, psychiatric and/or social reason)
2. Any clinically relevant gastrointestinal, renal, hepatic, neurological, haematological, endocrine, oncological, urological, immunological and cardiovascular diseases or any other condition including clinically significant abnormal laboratory parameters that, in the opinion of the Investigator, could jeopardise the safety of the subject or impact the validity of the study results
3. Lung cancer, upper respiratory tract cancers, chronic respiratory diseases or any other clinically significant pulmonary diseases according to the judgement of the Investigator
4. Any medical conditions requiring smoking cessation (e.g., recent acute cardiovascular event, diabetes mellitus, Chronic Obstructive Pulmonary disease)
5. Subject with body mass index < 18.5 or ≥ 30 kg/m2
6. As per judgement of the Investigator, medical conditions which require or will require in the course of the study a medical intervention (e.g., start of treatment, surgery, hospitalisation) which may interfere with the study participation and/or study results
7. Donation or receipt of whole blood or blood products within 3 months prior to the screening visit
8. Participation in any clinical studies within 3 months before the screening visit
9. Current or former employee of the tobacco industry, or of their first-degree relatives (parent, sibling, child)
10. Employee of the investigational site or any other parties involved in the study or of their first-degree relatives (parent, sibling, child)
11. Enrolled in the same study at a different time (i.e., each subject can be in the study population only once)
12. Subject who is legally incompetent, physically or mentality incapable of giving consent (e.g., emergency situation, under guardianship, subject in a social or sanitary establishment, prisoners or subject who are involuntarily incarcerated)
13. Positive alcohol test and/or history of alcohol abuse that could interfere with subject's participation in study
14. Positive urine drug tests (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates)
15. Positive serology test (HbsAg, HCV, HIV)

    Specific to smokers
16. Subject who has used any nicotine-containing products other than commercially available cigarettes (either a tobacco-based product or nicotine-replacement therapy) as well as electronic cigarettes and similar devices within 1 month prior to the screening visit

    Additionally, women of childbearing potential must be excluded if:
17. Subject is pregnant (does not have negative pregnancy tests at screening and at admission) or breastfeeding
18. Subject does not agree to use an acceptable method of effective contraception: intrauterine device, intrauterine system, established use of oral/injectable/implantable/transdermal hormonal methods, barrier methods of contraception (condoms, occlusive caps) with spermicidal foam/gel/film/suppository, vasectomised partner or true abstinence (periodic abstinence and withdrawal are not effective methods) from screening until the end of the safety follow-up period

Ages: 23 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Levels of CEMA, a biomarker of exposure to acrylonitrile, in 24-hour urine of smokers smoking 2 or 4 conventional cigarettes | After smoking 2 or 4 conventional cigarettes, within 24 hours
  To demonstrate that CEMA, used as a urinary biomarker, can identify subjects who have smoked 4 or less conventional cigarettes

SECONDARY OUTCOMES:
Levels of CEMA in 24-hour urine, carboxyhaemoglobin (COHb) in blood and carbon monoxide in exhaled breath of smokers smoking 2 or 4 conventional cigarettes | After smoking 2 or 4 conventional cigarettes, within 24 hours
  To evaluate the ability of CEMA to detect conventional cigarette use in comparison to COHb and exhaled carbon monoxide
Levels of CEMA, a biomarker of exposure to acrylonitrile, in 24-hour and spot urine of non-smokers | 24 hours
  To evaluate the correlation between the levels of CEMA in 24-hour urine and in spot urine in non-smokers

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Febbraro, MD, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, South Wales, United Kingdom